CLINICAL TRIAL: NCT03013335
Title: A Phase II Safety Trial of Nivolumab in Patients With Metastatic Renal Cell Carcinoma Who Have Progresses During or After Prior Systemic Anti-angiogenic Regimen
Brief Title: Nivolumab in Patients With Metastatic Renal Cell Carcinoma Who Have Progresses During or After Prior Systemic Anti-angiogenic Regimen
Acronym: NIVOREN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0160/1506 GETUG-AFU 26
Record Dates: First submitted 2016-11-10; First posted 2017-01-06 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Clear-cell; Nivolumab; Renal cell carcinoma; Immunotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab (Experimental): The dose and schedule of nivolumab in this study will be 3 mg/kg every 2 weeks. Infusion of nivolumab will be performed in 30 minutes (± 5 minutes).
  Nivolumab will be administered every 2 weeks until death, disease progression, unacceptable toxicity or withdrawal of the informed consent
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — The dose and schedule of nivolumab in this study will be 3 mg/kg every 2 weeks. Infusion of nivolumab will be performed in 30 minutes (± 5 minutes).
  Nivolumab will be administered every 2 weeks until death, disease progression, unacceptable toxicity or withdrawal of the informed consent

SUMMARY:
The primary objective of this study is to evaluate the incidence of high-grade (i.e. Grade 3-4 and Grade 5 of CTCAE v4.0) adverse reactions of interest in patients with metastatic RCC who have progressed during or after receiving at least one prior systemic anti-angiogenic treatment and who are eligible for nivolumab monotherapy.

DETAILED DESCRIPTION:
The present study will be carried out in patients suffering from refractory metastatic Renal Cell Carcinoma. The overall study population consists of 450 adult patients.

In France, 10600 patients were diagnosed with kidney cancer in 2010. At the time of their diagnosis, approximately 30% of patients present with metastatic disease, with 90 to 95% of that metastatic disease being of the clear-cell histology.

The present study is a multicenter, open-label, non-controlled, phase II safety study in patients who are suffering from metastatic Renal Cell Carcinoma and who have progressed during or after one prior systemic anti-angiogenic treatment. Patients intolerant to prior systemic anti-angiogenic treatment can also be eligible.

The dose and schedule of nivolumab in this study will be 3 mg/kg every 2 weeks. Nivolumab will be administered every 2 weeks until death, disease progression, unacceptable toxicity or withdrawal of the informed consent. 450 patients should be included over a period of 1 year

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women ≥18 years.
2. Patients with a histologically confirmed Renal Cell Carcinoma with a clear-cell component.
3. Patients with metastatic (AJCC stage IV) Renal Cell Carcinoma, with at least one measurable lesion by CT Scan or MRI according to RECIST 1.1 or with clinically apparent disease that can be reliably monitored by the investigator.
4. Patients having received at least one prior systemic anti-angiogenic treatment including but not limited to: sunitinib, sorafenib, pazopanib, axitinib, and bevacizumab, in the advanced or metastatic setting. Prior cytokine therapies (e.g. IL-2, IFN-α), vaccine therapy or treatment with cytotoxics are allowed. Patients intolerant to prior systemic anti-angiogenic treatment can also be eligible (except hypersensitivity to other monoclonal antibodies). A maximum of 25% of patients with more than 2 prior systemic treatments will be recruited per sites.
5. Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
6. Favorable, intermediate or poor risk group patients measured by the international metastatic renal cell carcinoma database consortium (IMDC) model.
7. Patients with brain metastases will be eligible if they are: asymptomatic, without edema, not on corticosteroids, not be eligible for radiation therapy/surgery and not receiving active treatments.
8. Patients who have progressed following radiation therapy. Palliative, focal radiation therapy, and immunosuppressive doses of systemic corticosteroids, except replacement organotherapy (hydrocortisone and fludrocortisone), must be discontinued at least 2 weeks prior to the first nivolumab administration.
9. Potentially reproductive patients must agree to use an effective contraceptive method or practice adequate methods of birth control or practice complete abstinence while on treatment, and for at least 31 weeks (≈ 7 months) for males and 23 weeks (≈ 5 months) for females after the last dose of study drug. Azoospermic males and women of childbearing potential who are continuously not heterosexually active are exempt from contraceptive requirements.
10. Women of childbearing potential must have a negative serum pregnancy test done within 24 hours prior to the first dosing.
11. Women who are breastfeeding should discontinue nursing prior to the first dose of study drug and until 6 months after the last dose.
12. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.
13. Patients with social insurance coverage.

Exclusion Criteria:

1. Patients with any active autoimmune disease or a history of known autoimmune disease (Patients with type I diabetes mellitus, residual hypothyroidism due to an autoimmune condition requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are however eligible for this trial).
2. Patients with uncontrolled adrenal insufficiency.
3. Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
4. Patients with positive tests for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection.
5. Patients having received prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
6. Patients having received any non-oncology vaccine therapy used for prevention of infectious diseases including seasonal (influenza) vaccinations within 4 weeks of the first dose of study drug.
7. Patients receiving anti-cancer therapies must be discontinued at least 2 weeks prior to administration of study drug. Palliative, focal radiation therapy, and immunosuppressive doses of systemic corticosteroids, except replacement organotherapy (hydrocortisone and fludrocortisone), must be discontinued at least 2 weeks before administration of study drug. All toxicities attributed to prior anti-cancer therapy other than alopecia must have resolved to grade 1 (NCI-CTCAE version 4) or baseline before administration of study drug.
8. Patients with other prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix or breast.
9. Patients with altered hematopoietic or organ function, as indicated by the following criteria (assessed within 14 days prior the first dosing):

   * White blood cell count <2000/µL
   * Polynuclear neutrophils <1.5 x 10⁹/L
   * Platelets <100 x 10⁹/L
   * Hemoglobin <8.0 g/mL
   * Alanine aminotransferase (ALAT)/ aspartate aminotransferase (ASAT) >3.0 x upper limit of normal (ULN) in the absence of liver metastases or >5 x ULN in the presence of liver metastases
   * Bilirubin >1.5 x ULN (except Gilbert Syndrome: <3.0 mg/dL)
   * Creatinine clearance ≤40 mL/min (measured or calculated by Cockcroft and Gault formula) or serum creatinine >2.0 x ULN
10. Patients with a history of hypersensitivity to other monoclonal antibodies or to the active or inactive excipients of study drug.
11. Known drug or alcohol abuse.
12. Known or underlying medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would make the administration of study drug hazardous to the patient or obscure the interpretation of toxicity determination or adverse events.
13. History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
14. Unwillingness to give written informed consent, unwillingness to participate, or inability to comply with the protocol for the duration of the study.
15. Individuals deprived of liberty or placed under the authority of a tutor.
16. Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to enrolment and during the treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence for high-grade (Grade3-4-5) adverse reactions of interest | 5 years
  The primary endpoint of this study is the incidence for high-grade (CTCAE v4.0 Grade 3-4 and Grade 5) adverse reactions of interest (i.e. adverse event related to study treatment).
  The adverse reactions of interest are: skin, endocrinopathy, gastrointestinal, hepatic, renal, pulmonary, and hypersensitivity adverse events.

SECONDARY OUTCOMES:
Assessment of Overall Survival (OS) by Follow-up continued | 5 years
  The efficacy data assessed by measuring the OS :
  OS is defined as the time from first dosing date to the date of death. A patient who has not died will be censored at last known date alive. OS will be followed continuously while patients are on the treatment and every 3 months via in-person or phone contact after patients discontinue the study drug.
Number of patients with a Best Overall Response (BOR) by RECIST v1.1 | 5 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 years
  Safety and tolerability will be measured by the incidence of all adverse events, serious adverse events, deaths and laboratory abnormalities. Adverse event assessments and laboratory tests will be performed at baseline, and continuously throughout the study at the beginning of each subsequent cycle.
Percentage of patients who received immune modulating concomitant medication | 5 years
  The percentage of patients who received immune modulating concomitant medication (e.g., corticosteroids, infliximab, cyclophosphamide, IVIG, mycophenolate mofetil), collected in a specific form.
Percentage of patients who received hormonal replacement therapy | 5 years
  The percentage of patients who received hormonal replacement therapy.
Median time to resolution of adverse reactions of interest | 5 years
  The median time to onset, median time to resolution (Grade 3-4) of adverse reactions of interest.
Assessment of quality of life by questionnaire FACT-G | 5 years
  Patient reported outcomes will be assessed by FACT-G
Assessment of quality of life by questionnaire FKSI-19 | 5 years
  Patient reported outcomes will be assessed by FKSI-19.
Assessment of quality of life by questionnaire EQ-5D | 5 years
  Global health status will be assessed by EQ-5D instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard ESCUDIER, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Laurence ALBIGES, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (7):
- France (7):
  - Centre Francois Baclesse, Caen
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy Cancer Campus Grand Paris, Villejuif

REFERENCES:
- [Derived] Rassy E, Dalban C, Colomba E, Derosa L, Alves Costa Silva C, Negrier S, Chevreau C, Gravis G, Oudard S, Laguerre B, Barthelemy P, Goupil MG, Geoffrois L, Rolland F, Thiery-Vuillemin A, Joly F, Ladoire S, Tantot F, Escudier B, Albiges L. Efficacy and Safety of Concomitant Proton Pump Inhibitor and Nivolumab in Renal Cell Carcinoma: Results of the GETUG-AFU 26 NIVOREN Multicenter Phase II Study. Clin Genitourin Cancer. 2022 Oct;20(5):488-494. doi: 10.1016/j.clgc.2022.07.003. Epub 2022 Jul 10. PMID 35977881
- [Derived] Billon E, Chanez B, Rochigneux P, Albiges L, Vicier C, Pignot G, Walz J, Chretien AS, Gravis G, Olive D. Soluble BTN2A1 Is a Potential Prognosis Biomarker in Pre-Treated Advanced Renal Cell Carcinoma. Front Immunol. 2021 Apr 20;12:670827. doi: 10.3389/fimmu.2021.670827. eCollection 2021. PMID 33959132
- [Derived] Flippot R, Dalban C, Laguerre B, Borchiellini D, Gravis G, Negrier S, Chevreau C, Joly F, Geoffrois L, Ladoire S, Mahammedi H, Rolland F, Gross-Goupil M, Deluche E, Priou F, Laramas M, Barthelemy P, Narciso B, Houede N, Culine S, Oudard S, Chenot M, Tantot F, Chabaud S, Escudier B, Albiges L. Safety and Efficacy of Nivolumab in Brain Metastases From Renal Cell Carcinoma: Results of the GETUG-AFU 26 NIVOREN Multicenter Phase II Study. J Clin Oncol. 2019 Aug 10;37(23):2008-2016. doi: 10.1200/JCO.18.02218. Epub 2019 Jun 13. PMID 31194611